CLINICAL TRIAL: NCT05767528
Title: Clinical Study of Neoadjuvant Therapy Outcome Prediction of Muscle-invasive Bladder Cancer Based on PTC Drug Sensitivity Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing GeneX Health Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Shaoxi Niu, Chinese People's Liberation Army (PLA) General Hospital, Chinese PLA General Hospital
Other Study IDs: S2022-714-01
Record Dates: First submitted 2023-02-15; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: Muscle-Invasive Bladder Carcinoma (MIBC); Patient-derived tumor-like cell clusters (PTC)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Case Group: Participants who were diagnosed as MIBC and plan to receive neoadjuvant therapy before the surgery, above 18 years of age, regardless of gender
  Interventions: Diagnostic Test: Patient-derived tumor-like cell clusters (PTC) drug sensitivity testing

INTERVENTIONS:
Diagnostic Test: Patient-derived tumor-like cell clusters (PTC) drug sensitivity testing — Conducting the neoadjuvant therapy of FDA-approved drugs for patients with muscle-invasive bladder carcinoma, culturing the patient-derived tumor-like cell clusters for drug sensitivity testing simultaneously, then assess the accuracy of the diagnostic test by combination and analysis of these results

SUMMARY:
In this study, investigators plan to conduct the 3D in vitro culture PTC drug sensitivity testing of fresh tumor specimen which obtained by endoscopic biopsy or other methods. Through assessing the consistency between the testing results and the patients' neoadjuvant treatment outcomes, they would evaluate the accuracy of PTC drug sensitivity testing and its application value in the individualized precision medicine for muscle-invasive bladder carcinoma.

DETAILED DESCRIPTION:
This is a prospective observational study. In this study, researchers propose to enroll 40 participants above 18 years of age with muscle-invasive bladder carcinoma, who are going to receive the neoadjuvant therapy before surgery. Collecting fresh tumor samples for PTC drug sensitivity testing, conducting neoadjuvant therapy for the subjects simultaneously. By combining PTC prediction results with the patients' clinical treatment process and medication feedback, researchers could estimate the accuracy of PTC drug sensitivity testing. Completion of this research would provide real-world figures to support for the clinical application for PTC drug sensitivity testing, and a method is going to be established to guide the clinical treatment regimen for patients with muscle-invasive bladder carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1 The lesion of biopsy was diagnosed as muscle-invasive bladder cancer
* 2 Age ≥ 18 years old, regardless of gender
* 3 Treatment plan of bladder removal surgery
* 4 Neoadjuvant therapy before surgery
* 5 Adequate fresh tumor tissue can be obtained by endoscopic biopsy for PTC drug sensitivity testing
* 6 ECOG 0-1, expected survival is more than 3 months
* 7 Normal or stable hepatic, renal, and hematopoietic function
* 8 Normal or stable blood pressure
* 9 The subjects are willing to participate, sign an informed consent form, and have good compliance

Exclusion Criteria:

* 1 Patients with incomplete clinical data
* 2 Central nervous system metastasis
* 3 The presence of other malignant diseases was discovered during treatment, which is going to interfere the study
* 4 Researchers believe that the patient is not suitable for participation after comprehensive evaluation
* 5 Refuse the treatment or follow-up plans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology patients with muscle-invasive bladder carcinoma above 18 years of age, at Chinese PLA General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | 3 months
  Disappearance of all target lesions. Any pathological lymph nodes（whether target or non-target）must have reduction in short axis to <10 mm. Length is measured in millimeters, refers to RECIST 1.1.
Partial Response (PR) | 3 months
  At least a 30％ decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Length is measured in millimeters, refers to RECIST 1.1.
Progressive Disease (PD) | 3 months
  At least a 20％ increase in the sum of diameters of target lesions, taking as reference the smallest sum on study（this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20％, the sum must also demonstrate an absolute increase of at least 5 mm.（the appearance of one or more new lesions is also considered progression). Length is measured in millimeters, refers to RECIST 1.1.
Stable Disease (SD) | 3 months
  Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Length is measured in millimeters, refers to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, M.D.&Ph.D., Principal Investigator — Chinese PLA General Hospital; Hongzhao Li, M.D.&Ph.D., Principal Investigator — Chinese PLA General Hospital; Shaoxi Niu, M.D.&Ph.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin S, Xi R, Wu A, Wang S, Li Y, Wang C, Tang L, Xia Y, Yang D, Li J, Ye B, Yu Y, Wang J, Zhang H, Ren F, Zhang Y, Shen D, Wang L, Ying X, Li Z, Bu Z, Ji X, Gao X, Jia Y, Jia Z, Li N, Li Z, Ji JF, Xi JJ. Patient-derived tumor-like cell clusters for drug testing in cancer therapy. Sci Transl Med. 2020 Jun 24;12(549):eaaz1723. doi: 10.1126/scitranslmed.aaz1723. PMID 32581131
- [Background] Feng RM, Zong YN, Cao SM, Xu RH. Current cancer situation in China: good or bad news from the 2018 Global Cancer Statistics? Cancer Commun (Lond). 2019 Apr 29;39(1):22. doi: 10.1186/s40880-019-0368-6. PMID 31030667
- [Background] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- [Background] Hoadley KA, Yau C, Wolf DM, Cherniack AD, Tamborero D, Ng S, Leiserson MDM, Niu B, McLellan MD, Uzunangelov V, Zhang J, Kandoth C, Akbani R, Shen H, Omberg L, Chu A, Margolin AA, Van't Veer LJ, Lopez-Bigas N, Laird PW, Raphael BJ, Ding L, Robertson AG, Byers LA, Mills GB, Weinstein JN, Van Waes C, Chen Z, Collisson EA; Cancer Genome Atlas Research Network; Benz CC, Perou CM, Stuart JM. Multiplatform analysis of 12 cancer types reveals molecular classification within and across tissues of origin. Cell. 2014 Aug 14;158(4):929-944. doi: 10.1016/j.cell.2014.06.049. Epub 2014 Aug 7. PMID 25109877
- [Background] Ciriello G, Miller ML, Aksoy BA, Senbabaoglu Y, Schultz N, Sander C. Emerging landscape of oncogenic signatures across human cancers. Nat Genet. 2013 Oct;45(10):1127-33. doi: 10.1038/ng.2762. PMID 24071851
- [Background] Wheler J, Lee JJ, Kurzrock R. Unique molecular landscapes in cancer: implications for individualized, curated drug combinations. Cancer Res. 2014 Dec 15;74(24):7181-4. doi: 10.1158/0008-5472.CAN-14-2329. Epub 2014 Oct 17. PMID 25326492
- [Background] Von Hoff DD, Stephenson JJ Jr, Rosen P, Loesch DM, Borad MJ, Anthony S, Jameson G, Brown S, Cantafio N, Richards DA, Fitch TR, Wasserman E, Fernandez C, Green S, Sutherland W, Bittner M, Alarcon A, Mallery D, Penny R. Pilot study using molecular profiling of patients' tumors to find potential targets and select treatments for their refractory cancers. J Clin Oncol. 2010 Nov 20;28(33):4877-83. doi: 10.1200/JCO.2009.26.5983. Epub 2010 Oct 4. PMID 20921468
- [Background] Tsimberidou AM, Iskander NG, Hong DS, Wheler JJ, Falchook GS, Fu S, Piha-Paul S, Naing A, Janku F, Luthra R, Ye Y, Wen S, Berry D, Kurzrock R. Personalized medicine in a phase I clinical trials program: the MD Anderson Cancer Center initiative. Clin Cancer Res. 2012 Nov 15;18(22):6373-83. doi: 10.1158/1078-0432.CCR-12-1627. Epub 2012 Sep 10. PMID 22966018
- [Background] Schwaederle M, Parker BA, Schwab RB, Daniels GA, Piccioni DE, Kesari S, Helsten TL, Bazhenova LA, Romero J, Fanta PT, Lippman SM, Kurzrock R. Precision Oncology: The UC San Diego Moores Cancer Center PREDICT Experience. Mol Cancer Ther. 2016 Apr;15(4):743-52. doi: 10.1158/1535-7163.MCT-15-0795. Epub 2016 Feb 12. PMID 26873727
- [Background] Le Tourneau C, Delord JP, Goncalves A, Gavoille C, Dubot C, Isambert N, Campone M, Tredan O, Massiani MA, Mauborgne C, Armanet S, Servant N, Bieche I, Bernard V, Gentien D, Jezequel P, Attignon V, Boyault S, Vincent-Salomon A, Servois V, Sablin MP, Kamal M, Paoletti X; SHIVA investigators. Molecularly targeted therapy based on tumour molecular profiling versus conventional therapy for advanced cancer (SHIVA): a multicentre, open-label, proof-of-concept, randomised, controlled phase 2 trial. Lancet Oncol. 2015 Oct;16(13):1324-34. doi: 10.1016/S1470-2045(15)00188-6. Epub 2015 Sep 3. PMID 26342236
- [Background] Prasad V. Perspective: The precision-oncology illusion. Nature. 2016 Sep 8;537(7619):S63. doi: 10.1038/537S63a. No abstract available. PMID 27602743
- [Background] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868
- [Background] Amendola LM, Jarvik GP, Leo MC, McLaughlin HM, Akkari Y, Amaral MD, Berg JS, Biswas S, Bowling KM, Conlin LK, Cooper GM, Dorschner MO, Dulik MC, Ghazani AA, Ghosh R, Green RC, Hart R, Horton C, Johnston JJ, Lebo MS, Milosavljevic A, Ou J, Pak CM, Patel RY, Punj S, Richards CS, Salama J, Strande NT, Yang Y, Plon SE, Biesecker LG, Rehm HL. Performance of ACMG-AMP Variant-Interpretation Guidelines among Nine Laboratories in the Clinical Sequencing Exploratory Research Consortium. Am J Hum Genet. 2016 Jun 2;98(6):1067-1076. doi: 10.1016/j.ajhg.2016.03.024. Epub 2016 May 12. PMID 27181684
- [Background] Sevin BU, Peng ZL, Perras JP, Ganjei P, Penalver M, Averette HE. Application of an ATP-bioluminescence assay in human tumor chemosensitivity testing. Gynecol Oncol. 1988 Sep;31(1):191-204. doi: 10.1016/0090-8258(88)90293-4. PMID 3410347
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484